CLINICAL TRIAL: NCT06034522
Title: A Single-Arm, Prospective, Clinical Investigation Evaluating the Safety and Feasibility of Adipearl Implantation in the Face of Adult Subjects
Brief Title: Clinical Investigation Evaluating the Safety and Feasibility of Adipearl
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Volumina Medical S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC0478
Record Dates: First submitted 2023-08-21; First posted 2023-09-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Mid-face Volume Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Face correction with Investigational device (Experimental): Subjects will be injected with the investigational device in the face.
  Interventions: Device: Adipearl

INTERVENTIONS:
Device: Adipearl — Injection of the investigational device in the face.

SUMMARY:
Adipearl is an injectable filler intended to be injected subcutaneously in the face.

ELIGIBILITY:
Inclusion Criteria:

* Subject having given freely and expressly informed consent;
* Subject deemed by the Investigator to be medically fit for injection of the product;
* Female or male subjects aged 22 to 65 years (inclusive);

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject participating to another research study.
* Subject with the presence of any condition, which in the opinion of the Principal Investigator, that makes her/him unable to complete the study per protocol.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Safety of Investigational Medical Device | Up to 6 months
  Collection of Injection Site Reactions and Adverse Events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Art Clinic, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No